CLINICAL TRIAL: NCT04619433
Title: A Multi-center, Randomized, Double-blind, Phase III Trial of SHR-1210 in Combination With Famitinib or Placebo Plus Chemotherapy in Subjects With Non-squamous Non-small-cell Lung Cancer.
Brief Title: A Study to Evaluate SHR-1210 in Combination With Famitinib Plus Chemotherapy in Subjects With NSCLC.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated by Sponsor
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1210-III-324
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Non-squamous Non-small-cell Lung Cancer
MeSH Terms: interventions — Carboplatin; famitinib; camrelizumab

STUDY DESIGN:
Intervention Model Description: SHR-1210 in combination with Famitinib plus chemotherapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A (Experimental): Intervention Drug: Camrelizumab; Pemetrexed; Carboplatin; Famitinib
  Interventions: Drug: Camrelizumab;Pemetrexed and Carboplatin; Famitinib;
- Treatment group B (Placebo Comparator): Intervention Drug: Camrelizumab; Pemetrexed; Carboplatin; Placebo
  Interventions: Drug: Camrelizumab;Pemetrexed and Carboplatin;Placebo

INTERVENTIONS:
Drug: Camrelizumab;Pemetrexed and Carboplatin; Famitinib; — Part 1:
  Drug: Camrelizumab; Pemetrexed; Carboplatin; Famitinib
  Part 2:
  Drug: Camrelizumab; Pemetrexed; Carboplatin; Famitinib
  Other Names: SHR1210
  Arms: Treatment group A
Drug: Camrelizumab;Pemetrexed and Carboplatin;Placebo — Part 2:
  Drug: Camrelizumab; Pemetrexed; Carboplatin; Placebo
  Other Names: SHR1210
  Arms: Treatment group B

SUMMARY:
The study is being conducted to evaluate the efficacy and safety of SHR-1210 in combination with Famitinib plus chemotherapy in subjects with NSCLC.

DETAILED DESCRIPTION:
The study is being conducted to evaluate the efficacy and safety of Camrelizumab in combination with Famitinib plus chemotherapy in subjects with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form, male or female, 18-70 years of age.
2. Histologically or cytologically confirmed, Stage IIIB-IV non-squamous NSCLC
3. EGFR mutation and ALK rearrangement status must be negative.
4. No prior system chemotherapy for advanced/metastatic NSCLC.
5. Measurable diseaseas defined by RECIST v1.1.
6. ECOG performance status of 0 or 1.
7. Has a life expectancy of at least 3 months.
8. Adequater organ function.
9. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose, and be willing to use a recognized effective contraceptive measure during the study and within 3 months after the last dose of the study drug; Male subjects with partners of childbearing potential must either be surgically sterilized or agree to take effective contraceptive measures during the study and within 3 months after the last dose of the study drug.

Exclusion Criteria:

1、 Cancer-Specific Exclusions

1. Other histological types of non-small cell lung cancer.
2. Subjects with carcinomatous meningitis and spinal cord compression.
3. Subjects with untreated central nervous system (CNS) metastasis.
4. Subjects who can be treated with surgical resection or radical radiotherapy.
5. Subjects who previously received anti-PD-1(L1) or CTLA4 monoclonal antibody, VEGF or VEGFR signaling pathway single target/multiple target inhibitor or monoclonal antibodies.

2. Medical history and complications

1. Subjects with any active, known, or suspected autoimmune diseases.
2. Subjects who require systemic corticosteroids prednisone (> 10 mg/day or equivalent) or other immunosuppressants within 14 days prior to the first dose.
3. Subjects who received cancer vaccines or other immunostimulatory anti-cancer agents (interferon, interleukin, thymosin, or immune cell therapy) within 1 month prior to the first dose.
4. Subjects who received anti-cancer TCM within 14 days prior to the first dose.
5. Subjects who are in another clinical study or last participated (last dose) in a clinical study less than 4 weeks (or 5 half-lives of the study drug) from the first dose, whichever is shorter.
6. Subjects who are expected to require other forms of anti-cancer treatment during the study.
7. Subjects who received major surgery within 4 weeks prior to the first dose, non-thoracic radiation therapy > 30 Gy within 4 weeks prior to the first dose, thoracic radiation therapy > 30 Gy within 24 weeks prior to the first dose, or palliative radiation ≤ 30 Gy within 2 weeks prior to the first dose, and failed to recover from the toxicities and/or complications of these interventions to NCI-CTC AE Grade ≤ 1 (except for alopecia and fatigue). Palliative radiotherapy for symptomatic control is permitted, but must be completed within 2 weeks prior to starting the study treatment.
8. Subjects highly suspected of interstitial lung disease, or with conditions that may interfere with the testing or management of suspected treatment-related pulmonary toxicities, or other moderate to severe lung diseases that seriously affect pulmonary function.
9. Subjects with a history of malignant tumors.
10. Subjects with severe cardiovascular disease.
11. Subjectss with hypertension which cannot be well controlled by antihypertensives.
12. Subjects with clinically significant hemorrhage or clear bleeding tendency within 3 month prior to the first dose.
13. Events of arterial/venous thrombosis within 6 months prior to the first dose.
14. Subjects who require long-term anticoagulant therapy with warfarin or heparin.
15. Subjects who require long-term antiplatelet therapy.
16. Significant vascular invasions or a high possibility of significant vascular invasions that may cause bleeding as determined by the investigator during treatment.
17. Subjects with active pulmonary tuberculosis (TB).
18. Subjects with serious infection within 4 weeks prior to the first dose, including but not limited to infective complications, bacteremia, and severe pneumonia that require hospitalization.
19. Subjects who prepare to receive or have previously received tissue/organ transplants.
20. Gastrointestinal disorder or surgical history that may affect the swallowing, digestion, and absorption of the oral drug as determined by the investigator.
21. Subjects who plan to receive or have received live vaccines within 30 days prior to the first dose.
22. Subjects with uncontrolled cancer pain.

3. Physical examination and laboratory tests

1. Known history of human immunodeficiency virus (HIV) seropositive status or acquired immunodeficiency syndrome (AIDS).
2. Active hepatitis B virus or hepatitis C virus infection.
3. Subjects with uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage.

4. Allergies and adverse drug reactions

1. Severe allergic reactions to other monoclonal antibodies.
2. Allergy or intolerance during an infusion.
3. History of severe allergies to pemetrexed, carboplatin, or their premedications.

5. Subjects with mental illness, alcohol abuse, inability to quit smoking, and drug or substance abuse.

6. Based on the investigator's judgment, subjects with a history or current evidence of diseases, treatments, or laboratory abnormalities that may affect study results, interfere with study procedures, or are not in the best interests of the subjects, should be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-08-16 (Actual); Study Completion 2025-08-16 (Actual)

PRIMARY OUTCOMES:
Part 1：Serum concentrations of Camrelizumab | Cycle 2; each cycle is 21 days (up to 42 days)
Part 1：Plasma concentrations of Famitinib | Cycle 2; each cycle is 21 days (up to 42 days)
Part 1：Area Under the Plasma Concentration Versus Time Curve (AUC) of Famitinib. | Cycle 2; each cycle is 21 days (up to 42 days)
Part 1：Maximum Concentration (Cmax) of Famitinib. | Cycle 2; each cycle is 21 days (up to 42 days)
Part 1：Time to Maximum Concentration (Tmax) of Famitinib. | Cycle 2; each cycle is 21 days (up to 42 days)
Part 1：Half-life (t1/2 z) of Famitinib. | Cycle 2; each cycle is 21 days (up to 42 days)
Part 1：Apparent Clearance (CL/F) of Famitinib | Cycle 2; each cycle is 21 days (up to 42 days）
Part 1：Vz/F of Famitinib. | Cycle 2; each cycle is 21 days (up to 42 days)
Part 2: Progression-free Survival (PFS) as Assessed by BICR according to RECIST 1.1. | up to 24 months

SECONDARY OUTCOMES:
Part 1:Objective Response Rate (ORR) as Assessed by investigators | Cycle 2; each cycle is 21 days (up to 42 days)
Part 1:Duration of Response (DOR) as Assessed by investigators | Cycle 2; each cycle is 21 days (up to 42 days)
Part 1:Progression-free Survival (PFS) as Assessed by investigators | Cycle 2; each cycle is 21 days (up to 42 days)
Part 1:Overall Survival (OS). | Up to approximately 60 months
Part 2:Overall Survival (OS) | Up to approximately 60 months
Part 2:Progression-free Survival (PFS) as Assessed by investigators according to RECIST 1.1. | up to 24 months
Part 2:Objective Response Rate (ORR) as Assessed by investigators and BICR according to RECIST 1.1 | up to 24 months
Part 2:Duration of Response (DOR) as Assessed by investigators and BICR according to RECIST 1.1 | up to 24 months
Part 2:Disease Control Rate(DCR) as Assessed by investigators and BICR according to RECIST 1.1 | up to 24 months
Part 2:Number of Participants With Adverse Events and Serious Adverse Event as Assessed by CTCAE v5.0. | up to 24 months

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Beijing Cancer Hosipital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospita, Wuhan, Hubei
  - Shengjing Hospita of China Medical University, Shenyang, Liaoning
  - Shanghai Lung Hospital, Shanghai, Shanghai Municipality
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality